CLINICAL TRIAL: NCT05358717
Title: A Phase 2A, Randomized, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety and Efficacy of PTC518 in Subjects With Huntington's Disease
Brief Title: A Study to Evaluate the Safety and Efficacy of PTC518 in Participants With Huntington's Disease (HD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PTC518-CNS-002-HD; 2021-003852-18 (EudraCT Number)
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Huntington Disease
Keywords: Neurodegenerative disorder; Rare disease
MeSH Terms: conditions — Huntington Disease; Neurodegenerative Diseases; Rare Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PTC518 5 mg (Experimental): Participants will receive PTC518 5 milligrams (mg) tablets once daily orally for 12 months.
  Interventions: Drug: PTC518
- PTC518 10 mg (Experimental): Participants will receive PTC518 10 mg tablets once daily orally for 12 months.
  Interventions: Drug: PTC518
- PTC518 20 mg (Experimental): Participants will receive PTC518 20 mg tablets once daily orally for 12 months.
  Interventions: Drug: PTC518
- Placebo (Placebo Comparator): Participants will receive placebo matching to PTC518 tablets once daily orally for 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PTC518 — PTC518 will be administered per dose and schedule specified in the arm.
  Arms: PTC518 10 mg; PTC518 20 mg; PTC518 5 mg
Drug: Placebo — Placebo matching to PTC518 will be administered per schedule specified in the arm.
  Arms: Placebo

SUMMARY:
The primary goal of this study is to evaluate the safety and pharmacodynamic effects of PTC518 compared with placebo in participants with HD.

DETAILED DESCRIPTION:
Participants will first be randomized to Part A or Part B or Parts D or E in a 1:1 randomization ratio, depending on their Huntington's disease Integrated Staging System (HD-ISS) staging criteria and then to active treatment (PTC518 5 mg in Parts A and D and 10 mg in Parts B and E) or matching placebo within each part in a 2:1 ratio of active treatment to placebo. A Drug Safety Monitoring Board (DSMB) Charter will undertake an unblinded review of safety data from the 5 and 10 mg dosing groups and provide a recommendation on when Parts C and F (with a 20 mg active treatment arm) can be initiated. At that time, participants will be randomized to any study Part that is currently open for enrollment, and then to either active treatment or placebo (in a 2:1 ratio) within that Part.

Participants who complete this study and agree to participate in a long-term extension (LTE) study, will be enrolled in a separate LTE study PTC518-CNS-004-HD (NCT06254482).

ELIGIBILITY:
Key Inclusion Criteria:

* Genetically confirmed HD diagnosis with a cytosine-adenine-guanine (CAG) repeat length from 40 to 50, inclusive

Eligibility for HD-ISS Stage 2 Group (Parts A, B, and C):

* A Unified Huntington's Disease Rating Scale (UHDRS)-Independence Scale (IS) score of 100
* A UHDRS Total Functional Capacity (TFC) score of 13
* A score between 0.18 and 4.93 inclusive on the normed version of the HD prognostic index (PINHD)

Eligibility for HD-ISS Mild Stage 3 Group (Parts D, E, and F):

* A UHDRS Total Functional Capacity (TFC) score of 11 or 12, or a UHDRS TFC score of 13 with an UHDRS IS score of <100

Key Exclusion Criteria:

* Receipt of an experimental agent within 90 days or 5 half-lives prior to Screening or anytime over the duration of this study, ribonucleic acid (RNA)- or deoxyribonucleic acid (DNA)-targeted HD-specific investigational agents such as antisense oligonucleotides, cell transplantation, or any other experimental brain surgery
* Any history of gene therapy exposure for the treatment of HD
* Participation in an investigational study or investigational paradigm (such as exercise/physical activity, cognitive therapy, brain stimulation, etc) within 90 days prior to Screening or anytime over the duration of this study
* Any medical history of brain or spinal disease that would interfere with the lumbar puncture process safety assessments
* Any medical history or condition that would interfere with the ability to complete the protocol-specified assessments (for example, implanted shunt, conditions precluding magnetic resonance imaging [MRI] scans)
* Pregnancy, planning on becoming pregnant during the course of the study or within 6 months of end of treatment, or currently breastfeeding

Note: Other inclusion and exclusion criteria may apply.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (4):
  - University of California, San Diego, La Jolla, California
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas Health Science Center at Houston; McGovern Medical School, Houston, Texas
  - University of Washington Department of Neurology, Seattle, Washington
- Australia (2):
  - Monash Health, Clayton
  - Westmead Hospital, Sydney
- Medical University Innsbruck, Innsbruck, Austria
- The Ottawa Hospital, Parkinson's and Movement Disorders Clinic, Ottawa, Canada
- France (3):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Hôpital Universitaire de Marseille Hôpital de la Timone, Marseille
  - Brain and Spine Institute Paris, Paris
- Germany (4):
  - Charite University Medicine Berlin, Berlin
  - Ruhr-Univ. Bochum St. Joseph-Hospital, Bochum
  - George-Huntington-Institut, Münster
  - Ulm University, UKU, Dep. of Neurology, Ulm
- Italy (3):
  - Irccs Istituto Delle Scienze Neurologiche Di Bologna Uoc Clinica Neurologica, Bologna
  - IRCCS Carlo Besta Neurological Institutte, Milan
  - IRCCS Casa Sollievo della Sofferenza Research Hospital, San Giovanni Rotondo
- Leiden University Medical Center, Leiden, Netherlands
- University of Otago, New Zealand Brain Research Institute, Christchurch, New Zealand
- Spain (4):
  - Hospital Universitario Cruces, Barakaldo
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario Burgos, Burgos
  - Hospital Ramón y Cajal, Madrid
- United Kingdom (4):
  - The Barbery National Centre for Mental Health, Birmingham
  - Cardiff University Schools of Medicine and Biosciences, Cardiff
  - UCL Queen Square Institute of Neurology National Hospital for Neurology and Neurosurgery, London
  - Manchester University NHS Foundation Trust, Manchester

REFERENCES:
- [Derived] Estevez-Fraga C, Tabrizi SJ, Wild EJ. Huntington's Disease Clinical Trials Corner: March 2024. J Huntingtons Dis. 2024;13(1):1-14. doi: 10.3233/JHD-240017. PMID 38489195
- [Derived] Estevez-Fraga C, Tabrizi SJ, Wild EJ. Huntington's Disease Clinical Trials Corner: November 2022. J Huntingtons Dis. 2022;11(4):351-367. doi: 10.3233/JHD-229006. PMID 36463457

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to receive placebo, PTC518 5 milligrams (mg), or PTC518 10 mg. While the Independent Data Monitoring Committee authorized opening of the 20 mg dosing arm, the sponsor elected not to open PTC518 20 mg dosing arm for enrollment.
Groups:
- Placebo: Participants received placebo matched to PTC518 tablets once daily (QD) orally for 12 months.
- PTC518 5 mg: Participants received 5 mg tablet of PTC518 QD orally for 12 months.
- PTC518 10 mg: Participants received 10 mg tablet of PTC518 QD orally for 12 months.
Period: Overall Study
Arm/Group | Placebo | PTC518 5 mg | PTC518 10 mg
Started | 53 | 52 | 54
Received at Least 1 Dose of Study Drug | 53 | 52 | 54
Completed | 51 | 47 | 51
Not Completed | 2 | 5 | 3
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Death | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Study Paused by Sponsor in United States | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population included all randomized participants who took at least 1 dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PTC518 5 mg | PTC518 10 mg | Total
Number analyzed (Participants) | 53 | 52 | 54 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (9.59) | 49.2 (9.04) | 47.8 (9.10) | 48.5 (9.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 26 | 29 | 88
  Male | 20 | 26 | 25 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 1 | 6
  Not Hispanic or Latino | 51 | 49 | 53 | 153
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 52 | 47 | 52 | 151
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 2 | 7

OUTCOME MEASURES:

1. Secondary Outcome: Percent Change From Baseline in Caudate Volume as Assessed Via Volumetric Magnetic Resonance Imaging (vMRI) at Month 12
Description: LS mean and standard error (SE) were calculated using MMRM.
Time Frame: Baseline, Month 12
Population: ITT Population included all randomized participants who took at least 1 dose of the study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | PTC518 5 mg | PTC518 10 mg
Number analyzed (Participants) | 53 | 52 | 54
percent change | 4.42 (0.413) [lower limit 0.413] | 4.99 (0.413) [lower limit 0.413] | 5.74 (0.391) [lower limit 0.391]

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A TEAE was defined as an AE that had an onset date or date of worsening on or after the first dose of study drug. A summary of other non-serious AEs and all serious adverse events (SAEs), regardless of causality is located in the 'Reported AE section'.
Time Frame: Baseline up to Month 18
Population: Safety Population included all randomized participants who received at least 1 dose of the study drug, with participants grouped according to the treatment they received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PTC518 5 mg | PTC518 10 mg
Number analyzed (Participants) | 53 | 52 | 54
Participants | 46 | 43 | 49

3. Primary Outcome: Percent Change From Baseline in Geometric Mean Blood tHTT Protein at Month 3
Description: Least square (LS) mean and 95% confidence interval (CI) were calculated using mixed-model repeated measures (MMRM). The blood tHTT protein value was log-transformed before fitting the MMRM model. The LS means from MMRM model were back-transformed to present geometric mean percent changes.
Time Frame: Baseline, Month 3
Population: ITT Population included all randomized participants who took at least 1 dose of the study drug.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | PTC518 5 mg | PTC518 10 mg
Number analyzed (Participants) | 53 | 52 | 54
percent change | -1.40 (-7.25) [-7.25 to 4.82] | -17.36 (-22.36) [-22.36 to -12.05] | -28.67 (-32.74) [-32.74 to -24.36]
Statistical Analysis 1: Comparison: Placebo vs PTC518 5 mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -15.97, 95% CI 2-sided [-23.59 to -8.34]
Statistical Analysis 2: Comparison: Placebo vs PTC518 10 mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -27.28, 95% CI 2-sided [-34.45 to -20.10]

4. Secondary Outcome: Change From Baseline in Composite Unified Huntington's Disease Rating Scale (cUHDRS) Scores at Month 12
Description: cUHDRS includes the Total Functional Capacity (range, 0-13; higher score means better functioning), Total Motor Score (range, 0-124; higher score means worse motor severity), Symbol Digit Modality Test (range, 0-110, correctly paired numbers-symbols in 90 seconds; higher score means better cognitive performance), and Stroop Word Reading (range, 0-no max value, correctly read colour words in 45 seconds; higher score means better cognitive performance) scores. The total score for the cUHDRS ranges from approximately 3 to 18, where higher scores indicated better functioning. LS mean and SE were calculated using analysis of covariance (ANCOVA) model.
Time Frame: Baseline, Month 12
Population: ITT Population included all randomized participants who took at least 1 dose of the study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | PTC518 5 mg | PTC518 10 mg
Number analyzed (Participants) | 53 | 52 | 54
units on a scale | -0.64 (0.168) [lower limit 0.168] | -0.61 (0.176) [lower limit 0.176] | -0.92 (0.164) [lower limit 0.164]

5. Secondary Outcome: Percent Change From Baseline in Geometric Mean Blood tHTT Protein at Month 12
Description: LS mean and 95% CI were calculated using MMRM. The blood tHTT protein value was log-transformed before fitting the MMRM model. The LS means from MMRM model were back-transformed to present geometric mean percent changes.
Time Frame: Baseline, Month 12
Population: ITT Population included all randomized participants who took at least 1 dose of the study drug.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | PTC518 5 mg | PTC518 10 mg
Number analyzed (Participants) | 53 | 52 | 54
percent change | 8.19 (1.99) [1.99 to 14.76] | -14.18 (-19.25) [-19.25 to -8.79] | -28.44 (-32.45) [-32.45 to -24.18]

6. Secondary Outcome: Percent Change From Baseline in Cerebrospinal Fluid (CSF) Mutant Huntingtin Protein (mHTT) at Month 12
Description: LS mean and 95% CI were calculated using MMRM. The CSF mHTT protein value was log-transformed before fitting the MMRM model. The LS means from MMRM model were back-transformed to present geometric mean percent changes.
Time Frame: Baseline, Month 12
Population: ITT Population included all randomized participants who took at least 1 dose of the study drug.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | PTC518 5 mg | PTC518 10 mg
Number analyzed (Participants) | 53 | 52 | 54
percent change | -15.64 (-26.71) [-26.71 to -2.90] | -23.68 (-33.97) [-33.97 to -11.78] | -23.28 (-32.84) [-32.84 to -12.35]

7. Secondary Outcome: Percent Change From Baseline in Blood mHTT Protein at Month 12
Description: LS mean and 95% CI were calculated using MMRM. The blood mHTT protein value was log-transformed before fitting the MMRM model. The LS means from MMRM model were back-transformed to present geometric mean percent changes.
Time Frame: Baseline, Month 12
Population: ITT Population included all randomized participants who took at least 1 dose of the study drug.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | PTC518 5 mg | PTC518 10 mg
Number analyzed (Participants) | 53 | 52 | 54
percent change | 13.89 (6.33) [6.33 to 21.98] | -14.11 (-19.99) [-19.99 to -7.79] | -28.20 (-32.89) [-32.89 to -23.20]

ADVERSE EVENTS:
Time Frame: Baseline up to Month 18
Description: Safety Population included all randomized participants who received at least 1 dose of the study drug, with participants grouped according to the treatment they received.
Groups:
- Placebo: Participants received placebo matched to PTC518 tablets QD orally for 12 months.
Arm/Group | Placebo | PTC518 5 mg | PTC518 10 mg
All-Cause Mortality (participants affected / at risk) | 1/53 | 1/52 | 0/54
Serious Adverse Events (participants affected / at risk) | 4/53 | 1/52 | 2/54
Other Adverse Events (participants affected / at risk) | 32/53 | 34/52 | 41/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=53) | PTC518 5 mg (N=52) | PTC518 10 mg (N=54)
Bone marrow oedema (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Drowning (General disorders) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=53) | PTC518 5 mg (N=52) | PTC518 10 mg (N=54)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (5) | 5 (6)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (5) | 1 (5)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (3) | 3 (3)
Fatigue (General disorders) | 3 (3) | 3 (3) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 2 (2) | 4 (4)
Influenza (Infections and infestations) | 9 (12) | 7 (7) | 9 (12)
Nasopharyngitis (Infections and infestations) | 9 (14) | 6 (8) | 8 (15)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (4) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 5 (7) | 8 (10) | 11 (16)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 3 (4) | 5 (5) | 3 (6)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 9 (10) | 8 (12)
Dizziness (Nervous system disorders) | 1 (1) | 3 (4) | 2 (2)
Headache (Nervous system disorders) | 7 (9) | 8 (30) | 13 (19)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 3 (4)
Tension headache (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3)
Depressed mood (Psychiatric disorders) | 3 (3) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 5 (5)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2023-10-05): https://cdn.clinicaltrials.gov/large-docs/17/NCT05358717/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT05358717/SAP_001.pdf